CLINICAL TRIAL: NCT03978364
Title: An Randomized Controlled Study of Azacitidine Combined With Homoharringtonine Compared With Azacitidine for Patients With Int/High -Risk MDS and AML-MRC
Brief Title: A Study of Azacitidine for Patients With Int/High -Risk MDS and AML-MRC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, director of hematology, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongPH004
Record Dates: First submitted 2019-03-20; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Myelodysplastic Syndromes,Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- azacitidine (Experimental): azacitidine
  azacitidine 75mg/m2，iH，qd， d1-7
  Interventions: Drug: Azacitidine regimen
- azacitidine combined HHT (Active Comparator): azacitidine+HHT azacitidine 75mg/m2，iH，qd， d1-7 HHT 3mg/m2,ivdrip qd,d1-3
  Interventions: Drug: Azacitidine combined HHT

INTERVENTIONS:
Drug: Azacitidine combined HHT — Azacitidine 75mg/m2，iH，qd×7days，HHT，3mg/m2 ivdrip qd×3 days
  Other Names: Azacitidine+HHT
  Arms: azacitidine combined HHT
Drug: Azacitidine regimen — Azacitidine 75mg/m2，iH，qd×7days，28 days a cycle
  Other Names: Azacitidine group
  Arms: azacitidine

SUMMARY:
evaluate the clinical efficacy and safety of azacitidine combined with HAG regimen for patients with int/high -risk MDS and AML-MRC with less than 30% blasts compared with azacitidine

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) is a group of heterogeneous clonal diseases originating from hematopoietic stem cells. The most common types of acute myeloid leukemia (AML) are AML with myelodysplasia-related changes (AML-MRC) and AML-NOS. AML-MRC patients are usually with multilineage pathological hematopoiesis, previous history of MDS or MDS-related cytogenetic abnormalities. Compared with AML-NOS, AML-MRC patients are usually older, with poor prognosis of cytogenetic changes, low remission rate of chemotherapy, and worse overall prognosis. The treatment strategies mainly include demethylation drugs, chemotherapy and allogeneic hematopoietic stem cell transplantation. The main purpose of treatment is to delay disease progression, prolong survival, and even be cured.

Epigenetic changes such as DNA methylation and histone deacetylation have been considered to be involved in the occurrence and development of MDS. Demethylation drugs, such as 5-azacitidine (AZA) and 5-aza-2-deoxycytidine (decitabine), can inhibit DNA methyltransferase, reduce excessive methylation of tumor suppressor genes, promote cell differentiation and apoptosis, and play an anti-tumor role. Demethylation drugs are important therapy for MDS patients. Compared with supportive treatment, demethylation drugs can reduce the risk of AML progression and improve survival.

Therefore, we proposed this project in order to further clarify the role of azacytidine in therapy for high-risk and middle-risk MDS and AML-MRC patients, and evaluate its clinical efficacy, to explore the optimal azacytidine treatment strategies for high-risk and middle-risk MDS and AML-MRC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-75 years old, male or female;
2. Int/high risk MDS AND AML patients (non-AML-M3) diagnosed according to the 2008 World Health Organization (WHO) diagnosis of myeloid malignant disease;
3. The ECOG behavior status score is 0-3 points;
4. The expected survival time is ≥ 3 months;
5. Ability to understand and be willing to sign the informed consent form of this trial.

Exclusion Criteria:

1. In the past, allergy to the drug contained in the test protocol or to a drug similar to the chemical structure of the test drug;
2. There are serious active infections;
3. Patients with clinically significant QTc interval prolongation (male > 450ms, female > 470ms), ventricular tachycardia (VT), atrial fibrillation (AF), grade II or higher heart block, myocardial infarction (MI) Patients with coronary heart disease who have congestive heart failure (CHF) within 1 year and who are symptomatic for medical treatment;
4. Heart B-ultrasound shows patients with end-diastolic pericardial cavity dark area width ≥ 10mm;
5. Patients with active bleeding;
6. Patients with new diseases such as thrombosis, embolism and cerebral hemorrhage in the past six months;
7. Abnormal liver function (total bilirubin > 1.5 times the upper limit of normal value, 2.5 times the upper limit of ALT / AST > normal value or 5 times the upper limit of ALT / AST > normal value in patients with liver invasion), abnormal renal function (serum Creatinine > 1.5 times the upper limit of normal);
8. The investigator determined that it was not suitable for the participants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, MD, PhD, Principal Investigator — Department of Hematology, Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China